CLINICAL TRIAL: NCT01804413
Title: Effects of Pegvisomant-Priming With the Glucagon Stimulation Test in Assessing GH and Cortisol Reserve in Adults: a Randomized Proof-of-Concept Pilot Study
Brief Title: Pegvisomant With Glucagon Test to Assess for Adult Growth Hormone Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Kevin Yuen, Associate Professor of Endocrinology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB6961
Record Dates: First submitted 2013-02-18; First posted 2013-03-05 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Adults Growth Hormone Deficiency.
Keywords: Pegvisomant; Growth hormone; Cortisol; Glucagon; Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — pegvisomant; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegvisomant-glucagon test (Active Comparator): To compare the combined pegvisomant with the glucagon test to the insulin tolerance test and the glucagon test in diagnosing adult growth hormone and cortisol insufficiency.
  Interventions: Drug: Pegvisomant; Drug: Regular insulin
- Insulin tolerance test (Active Comparator): To compare the combined pegvisomant with the glucagon test to the insulin tolerance test and the glucagon test in diagnosing adult growth hormone and cortisol insufficiency.
  Interventions: Drug: Regular insulin

INTERVENTIONS:
Drug: Pegvisomant — Pegvisomant 1 mg/kg injection 3 days before the glucagon test.
  Other Names: Somavert.
  Arms: Pegvisomant-glucagon test
Drug: Regular insulin — 0.1-0.15 units/kg

SUMMARY:
Hypothesis:

Pegvisomant combined with the glucagon stimulation test (GST) can improve the accuracy of this test when used to diagnose adult GH and cortisol (steroid hormone)insufficiency.

Study aims:

Diagnosing GH and cortisol deficiency in adults requires a special test. At present, the insulin tolerance test (ITT) is considered the test of choice. However, this test is difficult to perform as it involves giving insulin through the veins to decrease blood sugars to very low levels, and this can be unpleasant, and cannot be performed in elderly adults and in those with a history of heart disease, seizure disorders or stroke. For this reason there is an urgent need for an alternative reliable test. At present, the GST is considered the alternative test to the ITT but its accuracy in obese patients and in those with diabetes remains unclear. Pegvisomant is a medication that can increase GH production in the body. The purpose of this study is to find out if combining pegvisomant with the GST can help improve the accuracy of this test so that it is comparable with the ITT in diagnosing adult GH and cortisol insufficiency.

Study design:

Subjects will be recruited from the Oregon Health & Science University Dynamic Endocrine Testing Unit. A written informed consent will be obtained and a screening interview will be carried out. During the screening interview, the study will be explained to the subject in detail. For women of child-bearing age, a pregnancy test will be performed. The subjects will then take part in three studies on separate days: (1) GST; (2) pegvisomant (1 mg/kg) injection into the abdomen 3 days before the glucagon stimulation test (ii) insulin tolerance test. For the GST, glucagon will be injected into the muscle and blood draws will be performed every 30 mins for 240 mins. For the insulin tolerance test, a blood draw will be performed and insulin will be given into the vein followed by blood draws every 15 mins for 120 mins. The data from all three studies will be analyzed in the study where the peak growth hormone and cortisol levels for all three tests will be compared. A questionnaire will be used at the end of the study for the subjects to rank the level of preference of the three tests. The data of the study will be analyzed using a computer statistical program where the identity of the subjects will be coded to maintain confidentiality.

DETAILED DESCRIPTION:
Background: The diagnosis of GH deficiency in adults is established by provocative testing of GH secretion. The insulin tolerance test (ITT) is widely regarded as the gold standard test for diagnosing adult GH deficiency despite concerns about its practicality, safety, reproducibility, and its contraindications in elderly adults, adults with seizures and patients with ischemic heart disease. The glucagon stimulation test (GST) has been proposed as the alternative to the ITT for the following reasons: 1) availability; 2) low cost and 3) safety. This test has been validated in the past as a reliable test in assessing the GH reserve in both adults and children. In addition, a number of studies have also shown that the GST is capable of stimulating not only GH but also ACTH release. However, the accuracy and reliability of the GST in assessing the hypothalamic-pituitary-adrenal (HPA) axis and GH reserve in obese and diabetic patients are still lacking.

Pegvisomant (PV) (Somavert®) is a GH receptor antagonist and is currently licensed by the FDA for the treatment of acromegaly. Physiological studies have demonstrated that acute high dose administration of PV can enhance endogenous GH stimulation. These data was more recently utilized by Radetti et al. to prime the L-DOPA test in assessing its reliability in the diagnostic work up of GH deficiency in short children. Using a PV dose of 1 mg/kg to prime the L-DOPA test in 21 short children, these investigators demonstrated an improvement in the reliability of the L-DOPA stimulation test in diagnosing GH deficiency with 10 out of the 18 (56%) children that initially failed the L-DOPA test successfully passed the L-DOPA test following PV-priming. These investigators postulate that PV-priming unmasked potentially false diagnoses of GH deficiency by exploiting the acute IGF-lowering effect and reducing the negative feedback of GH on the hypothalamus.

We therefore propose this proof-of-concept pilot study to investigate the potential of acute GH receptor blockade using PV to reduce false positive rates in adults undergoing GH testing with the GST. In addition, we plan to investigate the effects of PV on IGF-I bioactivity, as measured by the IGF-I kinase receptor activation (KIRA) assay (30).

Subjects: Ten subjects with suspected pituitary disease will be invited to participate in the study. Subjects will be screened for eligibility before enrollment into the study.

Intervention: After completing the GST, eligible subjects will be randomized to undergo either the PV-GST or the ITT. Subjects who are randomized to undergo the PV-GST first will then undergo the ITT, and vice versa, 4-6 weeks later. For the PV-GST, a blood test for serum IGF-I and IGF-I KIRA level will be measured and the patient will then receive PV at a dose of 1 mg/kg injected subcutaneously. The patient will then return in 3 days' time to undergo the GST. For this part of the test, subjects will receive glucagon administered intramuscularly at a dose of 1 mg if subject weighs 90 kg or less and 1.5 mg if subject weighs more than 90 kg.

Measurements: Blood samples for the measurement of glucose, IGF-I, IGF-I KIRA, GH and cortisol will be performed at various time-points for the GST, PV-GST and ITT

Specific Aims:

Primary aims: 1) To investigate the potential of acute GH receptor blockade priming with PV to glucagon (PV-GST test) on the characteristics of peak GH and cortisol levels; 2) To ascertain cut-point levels for GH and cortisol with the PV-GST in comparison to the ITT in defining GH and cortisol deficiency.

Secondary aims: 1) Correlation between peak GH and cortisol levels induced by the PV-GST and BMI; 2) Correlation between peak GH and cortisol levels induced by the PV-GST and fasting blood glucose levels; 3) Effects of PV on IGF-I bioactivity as determined by the IGF-I KIRA.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age 21 to 55 years
* Body weight 60 to 120 kg inclusive
* Stable weight and diet for at least 3 months prior to study entry

Exclusion Criteria:

* Poor IV access
* Known hypersensitivity to glucagon
* Inability or unwillingness to comply with study procedures
* Clinically significant cardiovascular or cerebrovascular disease
* Current active malignancy other than non-melanoma skin cancer
* Active acromegaly or Cushing's disease
* Pheochromocytoma
* Pregnancy
* Renal failure (serum creatinine > 2 mg/dl)
* Severe acute illness
* Uncontrolled hypertension (BP > 160/100 mmHg)
* Emotional/social instability likely to prejudice study completion
* Recurrent or severe unexplained hypoglycemia
* Known or suspected drug/alcohol abuse
* Patients with history of coronary artery disease, cerebrovascular disease, congestive heart failure, arrhythmias and seizure disorder that would be excluded from the ITT arm regardless of age
* Participation in another simultaneous medical investigation or trial

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Peak growth hormone and cortisol levels induced by the pegvisomant-glucagon test compared to those by the insulin tolerance test in assessing the growth hormone and cortisol reserve in adults suspected of adult growth hormone and cortisol deficiencies. | 9 weeks
  Presently, the insulin tolerance test (ITT) is regarded as the gold standard test in diagnosing adult GH deficiency but this test is difficult to perform in patients with diabetes mellitus, and contraindicated in the elderly, and in adults with seizures and ischemic heart disease. Glucagon test is the alternative test to the ITT but its accuracy and reliability is questionable in obesity and diabetes mellitus. Pegvisomant is a GH receptor blocker that increases GH secretion. When primed with glucagon, pegvisomant may enhance GH secretion by providing a stronger stimulus than glucagon alone. We plan to assess if by priming pegvisomant with glucagon will improve the accuracy of this test in diagnosing adult GH cortisol deficiency. Specifically, we will examine the characteristics of peak GH and cortisol levels, and ascertain the peak GH and cortisol levels in comparison to those generated using the ITT in diagnosing GH and cortisol deficiency.

SECONDARY OUTCOMES:
Correlation of peak GH and cortisol levels to BMI and fasting glucose, and effects of pegvisomant on IGF-I bioactivity. | 9 weeks
  We plan to assess the correlation between peak growth hormone and cortisol levels induced by the pegvisomant-glucagon test and BMI, fasting blood glucose levels, and evaluate the effects of pegvisomant on insulin-like growth factor-I bioactivity using the insulin-like growth factor-I kinase receptor activity assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Yuen KC, Biller BM, Molitch ME, Cook DM. Clinical review: Is lack of recombinant growth hormone (GH)-releasing hormone in the United States a setback or time to consider glucagon testing for adult GH deficiency? J Clin Endocrinol Metab. 2009 Aug;94(8):2702-7. doi: 10.1210/jc.2009-0299. Epub 2009 Jun 9. PMID 19509104
- [Background] Berg C, Meinel T, Lahner H, Yuece A, Mann K, Petersenn S. Diagnostic utility of the glucagon stimulation test in comparison to the insulin tolerance test in patients following pituitary surgery. Eur J Endocrinol. 2010 Mar;162(3):477-82. doi: 10.1530/EJE-09-0824. Epub 2009 Dec 8. PMID 19996199
- [Background] Conceicao FL, da Costa e Silva A, Leal Costa AJ, Vaisman M. Glucagon stimulation test for the diagnosis of GH deficiency in adults. J Endocrinol Invest. 2003 Nov;26(11):1065-70. doi: 10.1007/BF03345251. PMID 15008242
- [Background] Gomez JM, Espadero RM, Escobar-Jimenez F, Hawkins F, Pico A, Herrera-Pombo JL, Vilardell E, Duran A, Mesa J, Faure E, Sanmarti A. Growth hormone release after glucagon as a reliable test of growth hormone assessment in adults. Clin Endocrinol (Oxf). 2002 Mar;56(3):329-34. doi: 10.1046/j.1365-2265.2002.01472.x. PMID 11940044
- [Background] di Iorgi N, Napoli F, Allegri A, Secco A, Calandra E, Calcagno A, Frassinetti C, Ghezzi M, Ambrosini L, Parodi S, Gastaldi R, Loche S, Maghnie M. The accuracy of the glucagon test compared to the insulin tolerance test in the diagnosis of adrenal insufficiency in young children with growth hormone deficiency. J Clin Endocrinol Metab. 2010 May;95(5):2132-9. doi: 10.1210/jc.2009-2697. Epub 2010 Mar 29. PMID 20350939
- [Background] Veldhuis JD, Bidlingmaier M, Anderson SM, Wu Z, Strasburger CJ. Lowering total plasma insulin-like growth factor I concentrations by way of a novel, potent, and selective growth hormone (GH) receptor antagonist, pegvisomant (B2036-peg), augments the amplitude of GH secretory bursts and elevates basal/nonpulsatile GH release in healthy women and men. J Clin Endocrinol Metab. 2001 Jul;86(7):3304-10. doi: 10.1210/jcem.86.7.7656. PMID 11443205
- [Background] Veldhuis JD, Bidlingmaier M, Anderson SM, Evans WS, Wu Z, Strasburger CJ. Impact of experimental blockade of peripheral growth hormone (GH) receptors on the kinetics of endogenous and exogenous GH removal in healthy women and men. J Clin Endocrinol Metab. 2002 Dec;87(12):5737-45. doi: 10.1210/jc.2001-011885. PMID 12466380
- [Background] Radetti G, Wu Z, Elsedfy HH, El Kholy M, Bozzola M, Strasburger CJ. Pegvisomant-primed GH stimulation test. Clin Endocrinol (Oxf). 2008 Jun;68(6):951-6. doi: 10.1111/j.1365-2265.2007.03132.x. Epub 2007 Nov 19. PMID 18031320
- [Derived] Yuen KC, Frystyk J, Rhoads SA, Bidlingmaier M. Pegvisomant-primed glucagon stimulation test in assessing GH reserve and GH/IGF kinetics in adults suspected of GH deficiency. Pituitary. 2016 Feb;19(1):65-74. doi: 10.1007/s11102-015-0688-8. PMID 26496767